CLINICAL TRIAL: NCT03768310
Title: Phase I Study of the Administration of CD19 Chimeric Antigen Receptor Multivirus-Specific Cytotoxic T Lymphocytes for Prophylaxis or Therapy of Relapse of CD19 Positive Malignancies After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: CD19.CAR-multiVSTs for Patients With CD19+ B-ALL or NHL Undergoing Related Allogeneic HSCT (CARMA)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We decided to move on to another product and as a result will not be moving forward with this study.
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rayne Rouce, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-36578 CARMA
Record Dates: First submitted 2018-11-20; First posted 2018-12-07 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Non-hodgkin Lymphoma; Acute Lymphoblastic Leukemia
Keywords: ALL; NHL; hematopoietic stem cell transplantation (HSCT)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CD19.CAR-multiVST for Group A (Experimental): Group A: Patients with no evidence of disease after having a bone marrow transplant.
  T cells will be given at the specified dose on or after day 30 after the bone marrow transplant. Three dose levels will be studied in both groups of patients (Group A and Group B). The lowest dose level will be 2 x 10^7cells/m2 and the highest will be 10 x10^7cells/m2.
  Interventions: Biological: CD19.CAR-multiVST for Group A
- CD19.CAR-multiVST for Group B (Experimental): Group B: Patients with evidence of disease before bone marrow transplant OR have relapsed after bone marrow transplant.
  Patients in Group B will receive the T cells at the earliest feasible time point after the detection of disease, but no earlier than day 30 after the transplant. The three dose levels will be studied in both groups of patients (Group A and Group B). The lowest dose level will be 2 x 10^7cells/m2 and the highest will be 10 x10^7cells/m2.
  Interventions: Biological: CD19.CAR-multiVST for Group B

INTERVENTIONS:
Biological: CD19.CAR-multiVST for Group A — Patients will be evaluated in the clinic and a single dose of CD19.CAR-multiVSTs will be given by intravenous injection on or after 30 days of the transplant (between days 30 and 90). A time period of 6 weeks will constitute the time for clinical safety monitoring.
  Other Names: CAR T Cells
  Arms: CD19.CAR-multiVST for Group A
Biological: CD19.CAR-multiVST for Group B — Patients will be evaluated in the clinic and a single dose of CD19.CAR-multiVSTs will be given by intravenous injection on or after 30 days of the bone marrow transplant. A time period of 6 weeks will constitute the time for clinical safety monitoring. If patients with relapse after transplant or those with evidence of disease before bone marrow transplant have at least a partial response to the treatment or have stable disease, they will be eligible to receive up to 6 additional doses of T cells separated by a minimum of four weeks. Patients are eligible to receive additional doses only after they have completed the initial 6-week clinical safety monitoring period.
  Other Names: CAR T Cells
  Arms: CD19.CAR-multiVST for Group B

SUMMARY:
This study is for patients that are having a bone marrow or stem cell transplant for either a type of cancer of the blood called Leukemia or a cancer of the lymph nodes called Non-Hodgkin's Lymphoma (NHL). Although a transplant can cure leukemia or lymphoma, some people will relapse (return of the disease). In those who relapse, current treatment cures only a very small percentage. This study is being conducted to evaluate the safety of a new type of therapy that may help to decrease the risk of relapse or treat relapse after it has occurred.

The body has different ways of fighting infection and disease. This study combines two of those ways, antibodies and T cells. Antibodies are proteins that protect the body from bacterial and other diseases. T cells are infection-fighting blood cells that can kill other cells, including tumor cells. Antibodies and T cells have been used to treat patients with cancers; they have shown promise, but have not been strong enough to cure most patients.

The antibody used in this study is called anti-CD19. This antibody is attracted to cancer cells because of a substance on the outside of these cells called CD19. For this study, the anti-CD19 antibody has been changed so that instead of floating free in the blood it is now joined to T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor (also known as a CAR T cell). Although anti-CD19 antibodies or chimeric receptors can kill cancer cells, unfortunately they sometimes do not last long enough to destroy all of the cancer cells.

These CD19 chimeric receptor multivirus specific T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the biggest dose of chimeric T cells that is safe to administer, to determine what the side effects are, to see how long the T cells last and to evaluate whether this therapy might help prevent infections and relapse in people with CD19+ leukemia or lymphoma having a bone marrow transplant.

DETAILED DESCRIPTION:
First, a donor gave us blood to make CD19 chimeric receptor multivirus specific T cells in the laboratory. These cells are grown and frozen for the patient. To make these special T cells, they are first stimulated with proteins specific for the target 5 viruses, then grow them with stimulator cells. These stimulator cells are irradiated (exposed to X ray waves in the laboratory) so that they can no longer grow. The proteins help the T cells learn to see and attack cells infected with CMV, EBV, Adv, BKV and HHV-6 (the target 5 viruses).

To get the CD19 antibody to attach to the surface of the T cell, the antibody gene is inserted into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps us find the T cells in the blood after injection. Once a sufficient number of T cells are made, they are frozen and tested to make sure they kill CD19+ tumor cells and cells infected with CMV, EBV, Adv, BKV and HHV-6 in the laboratory. The investigators will also test the cells to make sure they don't kill other normal cells in the body. Once testing is completed the cells will be ready to give to the patient.

Because the patient will have received cells with a new gene in them, the patient will be followed for a total of 15 years to see if there are any long term side effects of gene transfer. Because this is what is called a dose-escalation study, the investigators will be testing 3 different doses of T cells to find out which dose is safe, and possibly beneficial. When patients enroll on this study, they will be assigned a dose of CD19 chimeric receptor multivirus specific T cells. The dose received depends on the number of patients who have been treated before the patient, and how well they tolerated the T cells.

Patients will be given an injection of cells into the vein through an IV line at the assigned dose. Before they receive the injection, they may be given a dose of diphenhydramine (Benadryl) and acetaminophen (Tylenol). The injection will take about 10 minutes. The investigators will follow the patient in the clinic after the injection for up to 4 hours. Alternatively, if the patient has a high level of leukemia or lymphoma in the body, the investigators may decide to monitor the patient in the hospital after the injection. Patients will be required to remain local for at least 3 weeks after the T cell injection. This will be discussed before the treatment. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

Medical tests before treatment- Patients will receive a series of standard medical tests including physical exam and blood tests to measure blood cells, kidney and liver function.

Medical tests during and after treatment- Patients will receive standard medical tests when they are getting the infusions and after including physical exams and blood tests to measure blood cells, kidney and liver function.

To learn more about the way the CD19 chimeric receptor multivirus specific T cells are working and how long they last in the body, extra blood will be drawn. This blood may be drawn from a central line (existing long-term IV) if the patient has one. On the day patients receive the cells, blood will be taken before the cells are given and 3 hours afterwards. Other blood will be drawn one week, 2 weeks, 4 weeks, 6 weeks and 8 weeks after the infusion, then at Months 3, 6, 9 and 12. Because patients have had a bone marrow transplant, the majority of these time points would require a blood draw to check the standard medical tests anyway. However, some of these time points may involve an extra trip to clinic and blood draw. Then blood will be drawn every 6 months for 4 years, then yearly for a total of 15 years (up to 30 blood collections). If patients receive the cells at a time when sensitive tests indicate relapse or a high risk of relapse, patients will have additional reviews and blood tests to monitor these tests and look for relapse.

Patients will receive supportive care for acute (short) or chronic (long-term) toxicity, including blood components or antibiotics, and other intervention as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CD19+ B-ALL or NHL undergoing related allogeneic HSCT, with no evidence of disease post-HSCT (Group A) OR minimal residual disease (MRD) at time of HSCT OR relapse post-HSCT (Group B).

   Morphologic relapse (for Group B) will be defined by accepted definitions in Section 5.6 of the full protocol, and measured by PCR positivity, specific cytogenetic abnormalities, an abnormal population on flow cytometry or increased blasts on bone marrow biopsy or in the peripheral blood.

   MRD will be defined as detection in blood or marrow of any of the following (at time of transplant or on post-transplant evaluation): a) Any leukemia specific marker (such as t(9:22) or t(4:11)) documented in the patient's leukemia cells pre-transplant on a post-transplant evaluation b) An immune globulin rearrangement known to be a disease marker for this patient c) A leukemia specific phenotype at a level of > 0.01%95, 96 d) Mixed donor chimerism.
2. Age ≤ 75 years old
3. Patients with life expectancy ≥ 12 weeks
4. Patients with a Karnofsky/Lansky score ≥ 60
5. Related Donor approved for stem cell transplant
6. Patient or parent/guardian capable of providing informed consent
7. Patients with bilirubin less than or equal to 2x upper limit of normal
8. AST less than or equal to 3x upper limit of normal
9. Creatinine ≤2x upper limit of normal for age
10. Hemoglobin >7.0 (can be a transfused value)
11. Pulse oximetry of >90% on room air
12. Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the CTL infusion. The male partner should use a condom.
13. Available stem cell donor-derived CD19-CAR transduced multi-virus-specific cytotoxic T lymphocytes with 15% expression of CD19-CAR determined by flow-cytometry and <10% cytotoxicity against patient or donor-derived (or other family member-derived) PHA blasts.

Exclusion Criteria:

1. Severe intercurrent infection: Patients with a concurrent bacterial infection must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic antifungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
2. Evidence of graft versus host disease >grade II
3. Pregnant or lactating
4. History of hypersensitivity reactions to murine protein-containing products.
5. Currently taking corticosteroids for therapy of GVHD at a dose of >0.5mg/kg prednisone equivalent.
6. CNS abnormalities: Presence of CNS-3 disease defined as detectable cerebrospinal blast cells in a sample of CSF with ≥ 5 WBCs per mm3; History or presence of any CNS disorder such as a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
7. Patients who have received donor lymphocyte infusion (DLI) within 28 days.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2040-08 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose-Limiting Toxicities (DLT) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | 6 weeks
  DLT will be defined as any of the following that is NOT (1) pre-existing, or (2) due to infection (for which patients with B-ALL, B-Lly, and B-NHL are predisposed), or (3) due to underlying malignancy, and that may, after consultation with the FDA when indicated, be considered possibly, probably, or definitely related to the study cellular products.
  * Any Grade 5 event
  * Non-hematologic DLT is any grade 3 or 4 non-hematologic toxicity that fails to return to Grade 2 within 72 hours
  * Grade 2 to 4 allergic reaction to T cell infusion
  * Hematologic DLT is defined as any Grade 4 hematologic toxicity that fails to return to Grade 2 or baseline (whichever is more severe) within 14 days or within 28 days for patients with evidence of bone marrow disease
  * Acute GvHD grades III-IV within 42 days of the last T cell infusion

SECONDARY OUTCOMES:
Overall response rate according to RECIST criteria. | 4-8 weeks
  Overall response rate is defined as the proportion of subjects with best overall response of complete response (CR) or partial response (PR) according to RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rayne H Rouce, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hosptial, Houston, Texas
  - Texas Children's Hospital, Houston, Texas